CLINICAL TRIAL: NCT06520202
Title: A PHASE II PROSPECTIVE RANDOMIZED CROSSOVER STUDY ASSESSING THE ACUTE SAFETY & EFFICACY OF RHPRG4 (450 µG/ML RECOMBINANT HUMAN PROTEOGLYCAN 4) COMPARED TO VEHICLE FOR THE TREATMENT OF SJÖGREN'S RELATED DRY EYE DISEASE
Brief Title: RHPRG4 FOR THE TREATMENT OF SJÖGREN'S RELATED DRY EYE DISEASE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Efficacy signal substantial enough to move to a larger sturdy
Sponsor: Lubris Bio Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RHPRG4-SJÖGREN'S-001
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Sjogren's Syndrome With Dry Eye

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment Group (Experimental)
  Interventions: Drug: rhPRG4 (450 µg/mL)
- Vehicle Group (Active Comparator)
  Interventions: Drug: Vehicle
- Crossover Group (Experimental)
  Interventions: Drug: rhPRG4 (450 µg/mL)

INTERVENTIONS:
Drug: rhPRG4 (450 µg/mL) — 1-2 drops of rhPRG4 450 µg/mL solution in both eyes
  Arms: Crossover Group; Treatment Group
Drug: Vehicle — Sterile isotonic aqueous solution for ocular administration containing 0.01% polysorbate 20.
  Arms: Vehicle Group

SUMMARY:
A 1-day, randomized (1:1) controlled, masked, pre-market study. Subjects with moderate to severe Sjögren's related Dry Eye Disease will be evaluated at 0, 5, 30 & 90 minutes post dose of either rhPRG4 (Treatment group) or vehicle (Crossover group). At 90 minutes, Crossover group subjects will be administered rhPRG4, then evaluated 5 & 30 minutes after rhPRG4 instillation (95 & 120 minutes from baseline). All subjects will self-report for the remainder of the day at 4 hours and 8 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18-75 years of age.
2. Subjects previously diagnosed with Sjögren's Syndrome
3. Subjects diagnosed with Sjögren's related Dry Eye Disease for at least 3 months (current use of artificial tears for the treatment of Dry Eye)
4. VAS Eye Dryness (100-point scale) score ≥ 45 mm;
5. Osmolarity ≥ 312 mOsm/L in the worst performing eye;
6. Only subjects who satisfy all Informed Consent requirements may be included in the study.

Exclusion Criteria:

Diagnosis and Main Criteria for Exclusion:

1. Evidence of an active ocular infection in either eye;
2. History or presence of ocular surface disorders not related to dry eye in either eye, including but not limited to significant conjunctivochalasis, SLK, limbal stem cell deficiency, allergic conjunctivitis, GPC, AKC, anterior basement membrane dystrophies, recurrent corneal erosion, neurotrophic keratitis, PCEDs, exposure keratitis and moderate to severe blepharitis;
3. History of any ocular surgery (including laser or refractive surgical procedures) in either eye within 30 days before study enrollment. Ocular surgery will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period;
4. Presence or history of any ocular or systemic disorder or condition that might significantly hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct of trial procedures (e.g. ocular trauma, progressive or degenerative corneal conditions, uveitis, systemic infection), or initiation or cessation any systemic drug during the study period that is known to induce dry eye disease;
5. Known hypersensitivity to one of the components of the study or procedural medications;
6. Participation in another clinical study at the same time as the present study or within 14 days of screening/baseline visit;
7. History of drug, medication or alcohol abuse or addiction;
8. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:
9. are currently pregnant or,
10. have a positive result on the urine pregnancy test at the Screening/Baseline Visit or,
11. intend to become pregnant during the entire course of and 30 days after the study treatment periods, or,
12. are breast-feeding or,
13. not willing to use highly effective birth control measures, such as: Hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods, during the entire course of and 30 days after the study treatment periods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
• To assess the efficacy of rhPRG4 using the average VAS score assessing subjects' eye dryness (Question: Rate the dryness of your eye; anchors: 0 = no discomfort, 100 = maximal discomfort) at 90 minutes | 90 minutes
• To assess the safety of rhPRG4 by observation of the severity of treatment-emergent adverse events | 90 minutes

SECONDARY OUTCOMES:
• To assess the efficacy of rhPRG4 using the average VAS score for dryness, foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia and total VAS | at 5 minutes, 30 minutes, 90 minutes, 4 & 8 hours
• To assess the efficacy of rhPRG4 using the minimum inter-eye non-invasive tear film breakup time (TBUT): min(OU) | 30 minutes, 90 minutes
• To assess the efficacy of rhPRG4 using maximum inter-eye tear osmolarity: max(OU) | 30 minutes, 90 minutes
• To assess the efficacy of rhPRG4 using a patient questionnaire | 90 minutes
• To assess the safety of rhPRG4 by observation of the Best Corrected Visual Acuity (BCVA) | 90 minutes
• To assess the safety of rhPRG4 by observation of signs evaluated by slit lamp examination (SLE) | 90 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Sydney Eye Hospital, Sydney, Australia

IPD SHARING:
Plan to Share IPD: Undecided